CLINICAL TRIAL: NCT04933435
Title: Phase II Non-Randomized Trial of Interventional Radiology Liver Directed Therapies and Hypofractionated Image-Guided Radiation Therapy in Veteran and Non-Veteran, Non-surgical Hepatocellular Carcinoma Patients
Brief Title: Interventional Radiology Liver Directed Therapies and Hypofractionated Image-Guided Radiation Therapy in Veteran and Non-Veteran, Non-surgical Hepatocellular Carcinoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00089525_1
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Radiology Liver Directed Therapies (ILDT) (Active Comparator): ILDT includes ablations such as microwave ablation and percutaneous local ablation and embolotherapies including bland embolization, chemoembolization and radioembolization.
  Interventions: Other: Quality of life questionnaires
- Hypofractionated Image-Guided Radiation Therapy (HIGRT) (Active Comparator): HIGRT is a non-invasive, outpatient procedure typically delivered in 3-10 fractions of radiation.
  Interventions: Other: Quality of life questionnaires

INTERVENTIONS:
Other: Quality of life questionnaires — European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (QLQ-C30) and Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep)

SUMMARY:
This is a research study to evaluate change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC C-30), from baseline to 1 month post treatment in two patient cohorts receiving Interventional Radiology Liver Directed Therapies or Hypofractionated Image-Guided Radiation Therapy.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed either by histology/pathology or Liver Imaging Reporting and Data System (LIRADs 5 per the ACR's LIRADs criteria 10) by CT or MRI
* Patient is 18 years or older
* ECOG Performance status of 0-2
* Child Pugh score A5, A6, B7 or B8 (see Appendix)
* Lesion ≤ 5cm in size
* ≤ 3 lesions in the liver to be treated on protocol
* Lesion amenable to treatment with both Interventional Radiology Liver Directed Therapies and HIGRT.

Exclusion Criteria:

* Child Pugh score B9 or Class C
* Fluctuating ascites
* Inability to complete baseline Quality of Life survey forms
* Concurrent administration of systemic therapy for hepatocellular carcinoma
* Prior liver radiation therapy is an exclusion unless subject participation is approved by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
change in quality of life in patient cohorts receiving either Interventional Radiology Liver Directed Therapies or Hypofractionated Image-Guided Radiation Therapy | baseline, 1 month, 3 months, 6 months
  as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC C-30) measured from not at all (better) to very much (worse)

SECONDARY OUTCOMES:
change in quality of life in patients receiving Interventional Radiology Liver Directed Therapies or HIGRT | baseline, 1 month, 3 months, 6 months
  as measured by the FACT-Hep survey questionnaire from not at all (better) to very much (worse)
number of patients with grade ≥2 acute toxicity that received Interventional Liver Directed Therapy | 90 days
number of patients with grade ≥2 acute toxicity that received Hypofractionated Image Guided Radiation Therapy | 90 days
total healthcare system cost associated with Interventional Radiology Liver Directed Therapies | 90 days
total healthcare system cost associated with Hypofractionated Liver Directed Therapy | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Durham Veterans Administration Health Care System (DVAHCS), Durham, North Carolina
  - Duke Cancer Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No